CLINICAL TRIAL: NCT04830397
Title: A Randomized Active-controlled Multi-site Double-masked Study to Evaluate the Safety and Tolerability of 3 Concentrations of QLS-101 Versus Timolol Maleate Preservative Free (PF) 0.5% Ophthalmic Solution in Subjects With Primary Open-angle Glaucoma or Ocular Hypertension
Brief Title: Study to Evaluate QLS-101 Compared to Timolol Maleate Eye Drops in Subjects With High Eye Pressure (Glaucoma or Ocular Hypertension).
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Qlaris Bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QC-201
Record Dates: First submitted 2021-03-30; First posted 2021-04-05 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Primary Open Angle Glaucoma; Ocular Hypertension
Keywords: elevated intraocular pressure
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Timolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- QLS-101 0.5% (Experimental)
  Interventions: Drug: QLS-101
- QLS-101 1% (Experimental)
  Interventions: Drug: QLS-101
- QLS-101 2% (Experimental)
  Interventions: Drug: QLS-101
- Timolol Maleate 0.5% preservative free ophthalmic solution (Active Comparator)
  Interventions: Drug: Timolol Maleate

INTERVENTIONS:
Drug: QLS-101 — Ophthalmic solution 1x daily
  Arms: QLS-101 0.5%; QLS-101 1%; QLS-101 2%
Drug: Timolol Maleate — Ophthalmic solution 1x daily
  Arms: Timolol Maleate 0.5% preservative free ophthalmic solution

SUMMARY:
Evaluating the safety and tolerability of QLS-101 versus timolol maleate ophthalmic solution in glaucoma or ocular hypertension.

DETAILED DESCRIPTION:
Multi-site study to evaluate the safety and tolerability of 3 concentrations of QLS-101 versus timolol maleate Preservative Free (PF) 0.5% ophthalmic solution in subjects with primary open-angle glaucoma or ocular hypertension

ELIGIBILITY:
Inclusion Criteria:

1. Visual acuity +1.0 logMAR or better
2. Willing to give informed consent
3. Ability to washout from current intraocular pressure lowering medications -

Exclusion Criteria:

1. Severe glaucomatous damage
2. Previous glaucoma intraocular or laser surgery
3. Refractive surgery
4. Ocular infection or inflammation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2021-03-31 (Actual); Primary Completion 2022-02-17 (Actual); Study Completion 2022-02-17 (Actual)

PRIMARY OUTCOMES:
Ocular safety | 100 days
  Number of participants with treatment-related adverse events will be monitored

SECONDARY OUTCOMES:
Ocular hypotensive efficacy | 28 days
  Number of participants with intraocular pressure reduction from baseline will be calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Dixon Eye Care, Albany, Georgia, United States

REFERENCES:
- See also: Company website, pipeline — https://qlaris.bio